CLINICAL TRIAL: NCT00000727
Title: A Controlled Comparative Trial of Trimethoprim - Sulfamethoxazole Versus Aerosolized Pentamidine for Secondary Prophylaxis of Pneumocystis Carinii Pneumonia in AIDS Patients Receiving Azidothymidine (AZT)
Brief Title: A Controlled Comparative Trial of Sulfamethoxazole-Trimethoprim Versus Aerosolized Pentamidine for Secondary Prophylaxis of Pneumocystis Carinii Pneumonia in AIDS Patients Receiving Azidothymidine (AZT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 021; 10997 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Sulfadoxine; Trimethoprim-Sulfamethoxazole Combination; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Pentamidine; Pyrimethamine; Drug Evaluation; Administration, Inhalation; Administration, Oral; Aerosols; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; AIDS-Related Opportunistic Infections; Respiratory Aspiration; Acquired Immunodeficiency Syndrome | interventions — Pentamidine; Pyrimethamine; Trimethoprim, Sulfamethoxazole Drug Combination; fanasil, pyrimethamine drug combination; Zidovudine

INTERVENTIONS:
Drug: Pentamidine isethionate
Drug: Pyrimethamine
Drug: Sulfamethoxazole/Trimethoprim
Drug: Sulfadoxine/Pyrimethamine
Drug: Zidovudine

SUMMARY:
To determine if the drug combination sulfamethoxazole-trimethoprim (SMX-TMP), given by mouth, and the drug pentamidine (PEN), given by inhaled aerosol, are effective in preventing a relapse of Pneumocystis carinii pneumonia (PCP) when they are given to patients who have recovered from a first episode of PCP and are being given zidovudine (AZT) to treat primary HIV infection.

AZT prolongs survival in patients with AIDS and decreases the occurrence of opportunistic infections such as PCP. However, PCP recurs in about 43 percent of patients receiving AZT, indicating a need for other treatments to reduce the relapse rate.

The two medications to be tested in this study, SMX/TMP and aerosolized PEN, have also been partially effective in preventing recurrence of PCP. It is hoped that the combination of AZT with these medications will be more effective than AZT or one of the medications alone.

DETAILED DESCRIPTION:
AZT prolongs survival in patients with AIDS and decreases the occurrence of opportunistic infections such as PCP. However, PCP recurs in about 43 percent of patients receiving AZT, indicating a need for other treatments to reduce the relapse rate.

The two medications to be tested in this study, SMX/TMP and aerosolized PEN, have also been partially effective in preventing recurrence of PCP. It is hoped that the combination of AZT with these medications will be more effective than AZT or one of the medications alone.

Patients receive the standard dose of AZT at study entry. Low body weight patients receive AZT at a lower dose. Patients are randomly assigned to one of two medications intended to prevent the recurrence of PCP. Patients assigned to SMX/TMP will take 1 capsule which contains both drugs once a day for 1 year. Patients assigned to PEN will have 1 aerosol treatment every 4 weeks for 1 year. Blood will be drawn at intervals in order to estimate blood levels of the drugs and to detect any adverse effects from the drugs. Note: Earlier versions of this protocol reflect its original design as a 3-arm study comparing aerosolized PEN, SMX/TMP, and pyrimethamine-sulfadoxine as secondary prophylaxis of PCP in AIDS patients receiving AZT. In order to reduce the effective sample size and permit the completion of accrual in a reasonable period of time, the pyrimethamine - sulfadoxine arm of this study has been discontinued. Patients randomized to this arm will be continued in this study on the original randomized therapy. Management of these patients will follow that described for SMX/TMP in the latest protocol version. AMENDED: Lower dose of AZT allowed.

ELIGIBILITY:
Inclusion Criteria

Patients must fulfill the following criteria:

* Randomization within 10 weeks of completing therapy for Pneumocystis carinii pneumonia (PCP).
* Ability to tolerate oral and aerosolized therapy at the time of randomization.
* Life expectancy > 4 months.

Concurrent Medication:

Allowed:

* Inhaled bronchodilators for cough and bronchospasm related to aerosolized pentamidine treatment.
* Aspirin at modest doses.
* Ibuprofen at modest doses.
* Acetaminophen at modest doses.
* Erythropoietin for management of anemia.
* Allowed to treat opportunistic infections while on study:
* Acyclovir.
* Ketoconazole.
* Amphotericin B.
* Nystatin.
* Clotrimazole.
* Also allowed:
* Ganciclovir (DHPG) for maintenance therapy of life-threatening or sight-threatening cytomegalovirus retinitis (CMV retinitis) infection only.
* Zidovudine (AZT) must be discontinued during the acute induction phase of treatment and will be restarted when maintenance therapy is introduced.

Concurrent Treatment:

Allowed:

* Local radiation therapy for Kaposi's sarcoma.

Prior Medication:

Allowed:

* Primary prophylactic therapy prior to Pneumocystis carinii pneumonia (PCP) episode.

Risk Behavior:

Allowed:

* Patients maintained in a methadone maintenance program per local investigator's judgment.

Exclusion Criteria

* Active drug or alcohol abuse which would impair performance as a study subject.

Concurrent Medication:

Excluded:

* Famotidine.
* Any medications suspected of interference with the metabolism of zidovudine.
* Flurazepam.
* Chronic probenecid.
* Phenobarbital.
* Phenytoin.
* Experimental therapies, except as noted.
* Chronic oral bronchodilators should not be started in patients in order to maintain them on aerosolized pentamidine after they have exhibited pulmonary toxicity.

Prior Medication:

Excluded for the 30 patients who will undergo pharmacokinetic studies:

* Zidovudine (AZT) at any time.
* Excluded within 7 days of study entry for the 30 patients who will undergo pharmacokinetic studies:
* Trimethoprim / sulfamethoxazole.
* Pyrimethamine / sulfadoxine.
* Aerosolized pentamidine.
* Excluded:
* Pentamidine by any route for the original infection.
* Prophylactic therapy for Pneumocystis carinii pneumonia (PCP) between the discontinuation of acute treatment and study entry.

Prior Treatment:

Excluded within 2 weeks of study entry:

* Transfusions of blood or red blood cells.

Patients may not have any of the following symptoms or diseases:

* Known treatment-limiting hypersensitivity to sulfonamides, trimethoprim, pyrimethamine, pentamidine, or zidovudine (AZT), especially but not limited to, exfoliative dermatitis, erythema multiforme, and Stevens-Johnson syndrome.
* Development of severe hypoglycemia (serum glucose < 50 mg/dl with pentamidine therapy).
* History of neoplasms other than basal cell carcinoma of the skin or carcinoma in situ of the cervix, or mucocutaneous Kaposi's sarcoma.
* Known visceral Kaposi's sarcoma.
* Known glucose-6-phosphate dehydrogenase (G-6-PD) deficiency.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322
Dates: Study Completion 1991-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holzman R, Study Chair; Hardy WD, Study Chair
Locations (9):
- United States (9):
  - USC CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Bmc Actg Crs, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Case CRS, Cleveland, Ohio
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Freedberg KA, Hardy WD, Holzman RS, Tosteson AN, Craven DE. Validating literature-based models with direct clinical trial results: the cost-effectiveness of secondary prophylaxis for PCP in AIDS patients. Med Decis Making. 1996 Jan-Mar;16(1):29-35. doi: 10.1177/0272989X9601600110. PMID 8717596
- [Background] Hardy WD, Feinberg J, Finkelstein DM, Power ME, He W, Kaczka C, Frame PT, Holmes M, Waskin H, Fass RJ, et al. A controlled trial of trimethoprim-sulfamethoxazole or aerosolized pentamidine for secondary prophylaxis of Pneumocystis carinii pneumonia in patients with the acquired immunodeficiency syndrome. AIDS Clinical Trials Group Protocol 021. N Engl J Med. 1992 Dec 24;327(26):1842-8. doi: 10.1056/NEJM199212243272604. PMID 1448121
- [Background] Hardy WD, Holzman RS, Avramis V, Bawdon R, Fall H, Feinberg J. Clinical and pharmacokinetic interactions of combined zidovudine (ZDV) therapy and sulfadoxine-pyrimethamine (fansidar) prophylaxis in post-PCP AIDS patients (ACTG 021). Int Conf AIDS. 1989 Jun 4-9;5:294 (abstract no TBP46)
- [Background] Robins JM, Finkelstein DM. Correcting for noncompliance and dependent censoring in an AIDS Clinical Trial with inverse probability of censoring weighted (IPCW) log-rank tests. Biometrics. 2000 Sep;56(3):779-88. doi: 10.1111/j.0006-341x.2000.00779.x. PMID 10985216